## A single center randomized prospective study on the criteria for lymph node sorting for pathological examination after curative surgery for gastric cancer

(DJY001 Trail)

**Edition Number: 1.0** 

**Edition Generation Date: Qct 30, 2017** 

Principal Investigator: Jingyu Deng and Han Liang

Research Institute: Cancer Hospital & Institute of Tianjin Medical University

## **Protocol:**

